CLINICAL TRIAL: NCT02454426
Title: An 8-week, Open-Label Clinical Trial of the Efficacy and Safety of Vortioxetine in Patients With Major Depressive Disorder and Coronary Artery Disease
Brief Title: Vortioxetine in Patients With Major Depressive Disorder and Coronary Artery Disease
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: PI left institution
Sponsor: Thomas Jefferson University (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TakedaHRV
Record Dates: First submitted 2015-05-21; First posted 2015-05-27 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: Major Depressive Disorder; Coronary Artery Disease
Keywords: Depression; Heart disease
MeSH Terms: conditions — Depressive Disorder, Major; Coronary Artery Disease; Depression; Heart Diseases | interventions — Vortioxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open-Label Treatment (Experimental): Patients will be initiated on vortioxetine 5 mg/day for 4 days, then increased to 10 mg/day. After the week 2 visit, patients will then be increased to 20 mg/day for the remainder of the study
  Interventions: Drug: Vortioxetine

INTERVENTIONS:
Drug: Vortioxetine — open label treatment
  Other Names: Brintellix

SUMMARY:
This is a preliminary, open-label, clinical trial designed to assess the efficacy, safety, and tolerability of vortioxetine for the treatment of major depressive disorder in patients with coronary artery disease. In addition, the study will assess the effects of vortioxetine on heart rate variability in these patients.

DETAILED DESCRIPTION:
Comorbid Major Depressive Disorder (MDD) and Coronary Artery Disease (CAD) are common:

Major depressive disorder is a highly prevalent disorder that is serious, and in some cases life-threatening, condition. The 12-month prevalence of major depressive disorder in the United States is 6.6% (Kessler et al., 2003). Coronary artery disease (CAD) is also a large and growing problem in the United States. According to the 2014 American Heart Association (AHA) report on heart disease and stroke statistics, an estimated 15.4 million Americans ≥20 years of age have coronary artery disease. The total prevalence of coronary artery disease in this population is estimated to be 6.4%, with a prevalence of 7.9% in men and 5.1% in women. By the year 2030, the prevalence of coronary artery disease is projected to increase approximately 18% from 2013 estimates (Go et al., 2014). Thus, patients with major depressive disorder and comorbid CAD represent a large population of patients.

Depression in patients with CAD is clinically important:

Depression frequently accompanies coronary artery disease and has been linked more somatic symptoms, hospitalizations, increased financial burden, and poorer quality of life, as well as being a predictor of worse outcomes of cardiac disease. Reduction of cardiac risk factors is less likely to be successful in depressed patients. Depression may also interfere with medication adherence, as depressed patients are three times as likely to be noncompliant with their medication regimens. In addition, depression is associated with decreased rates of participation in cardiac rehabilitation, higher healthcare utilization and costs, and greatly reduced quality of life (Lichtman et al., 2009). Due to these effects of depression on coronary artery disease, there is increasing recognition that depression should be formally considered a risk factor for adverse medical outcomes in patients with acute coronary syndrome (Lichtman et al., 2014).

Thus, there is a great, unmet clinical need to treat patients with major depressive disorder and coronary artery disease.

In addition to the older tricyclic antidepressants, the newer serotonin-norepinephrine reuptake inhibitors are also associated with cardiovascular risks like hypertension, orthostatic hypotension, and perhaps QTc prolongation (Mago et al., 2014). Vortioxetine is a newly approved antidepressant thought to work by combining modulation of 5-HT receptor subtypes and inhibition of the serotonin transporter (Citrome, 2014). Early data suggests that this multimodal mechanism of action results in increased brain levels of serotonin, dopamine, and noradrenaline in the prefrontal cortex (Pehrson et al., 2013). Clinical trials of vortioxetine for major depressive disorder have not shown any cardiovascular adverse effects (Mago et al., 2014).

Heart Rate Variability (HRV) Heart Rate Variability is a measure is based on the changes in the interval between consecutive heart beats and between consecutive instantaneous heart rates. It has become the conventionally accepted term to describe variations of both instantaneous heart rate and RR intervals. Long term reduced heart rate variability can lead to immune dysfunction and inflammation, cardiovascular disease and mortality (Newhouse, 2014). Several studies in depressive patients have shown reduced heart rate variability that suggests an increased sympathetic activity and/or reduced vagal activity (Carney et al., 2009). Thus, treating depression effectively may reduce heart rate variability, which is a surrogate marker for better cardiovascular outcomes.

The proposed study has been planned as a pilot, open-label study of the use, for the first time, of vortioxetine in patients with documented coronary disease. Therefore, the sample size is not based on a formal sample size calculation but on feasibility of a small study that, if positive, can lead to a future larger, adequately powered study. A sample size of 25 patients is appropriate for the present purpose. The results of this proposed study would inform sample size calculation for a future, larger study.

ELIGIBILITY:
Inclusion Criteria:

1. DSM-5 diagnosis of a major depressive disorder based on clinical evaluation by the study psychiatrist
2. At least moderate severity of depression as indicated by a Montgomery-Asberg Depression Rating Scale (MADRS) score of 22 or greater
3. History of coronary artery disease as defined by:

   * History of coronary stenosis in one or more vessels that is greater ≥ 70% by coronary angiography or CT angiogram, OR
   * History of abnormal stress test (at least medium-sized, moderate, reversible defect), OR
   * History of documented myocardial infarction including ST elevation myocardial infarction or non-ST elevation myocardial infarction (with elevated troponins), OR
4. Evidence of adequate treatment of the coronary artery disease as defined by at least one of the following that was done at least six months prior to the Screening visit, AND was followed by the patient being clinically stable in the opinion of a cardiologist who has evaluated the case:

   * Coronary artery bypass grafting (CABG)
   * Percutaneous coronary intervention (PCI)/ stenting
   * Adequate management with optimal medical treatment (such as one or more of the following medications: aspirin, beta blockers, a statin (e.g., atorvastatin), and either an ACE inhibitor or an angiotensin-receptor blocker.)

Key Exclusion Criteria:

Psychiatric Exclusion Criteria:

1. Patients who in the past have failed to respond to a trial of vortioxetine at the minimum recommended dose (10 mg/day) or greater taken for at least six weeks, or had unacceptable adverse effects while taking vortioxetine.
2. Patients must not have failed treatment with more than one antidepressant (taken at an adequate dose and for at least six weeks) in the current episode of major depressive disorder (i.e., did not have > 50% reduction in severity of depression based on patient history)
3. Patients with a current primary DSM-5 diagnosis of:

   i) Delirium, dementia, amnestic, or other cognitive disorder; ii) Eating Disorder (including Anorexia Nervosa or Bulimia); iii) Obsessive Compulsive Disorder; iv) Panic Disorder; v) Post-Traumatic Stress Disorder (PTSD);
4. Current or past (lifetime) DSM-5 diagnosis of:

   i) Bipolar I or II disorder; ii) Hypomanic episode iii) Substance-induced manic or hypomanic episode iii) Schizophrenia or other psychotic disorder

Cardiovascular Exclusion Criteria:

1. Patients who have had a myocardial infarction within 30 days of the screening visit
2. Any cardiovascular condition that is unstable or decompensated
3. In the opinion of the Investigators, the patient is at significant risk of cardiovascular adverse events
4. Coronary artery bypass grafting (CABG) or percutaneous coronary intervention (PCI)/ stenting within three months of the screening visit
5. Admission to a hospital for any cardiac condition within three months of the screening visit
6. Decompensated heart failure within 6 months of the screening visit
7. QTc prolongation (screening ECG with QTc ≥ 450 msec for men or QTc ≥ 470 msec for women) using QTc Fridericia correction
8. Second-degree (if Mobitz II) or third-degree atrioventricular block
9. Heart rate on ECG of ≤ 50 bpm or ≥ 120 bpm or any heart rate that is clinically symptomatic
10. Premature Ventricular Contractions (PVCs) associated with clinical symptoms and/or any complex premature ventricular contractions (ie, PVCs that are frequent [> 30/hr] or ≥ 2 beats if multifocal, or show bigeminy, trigeminy, quadrigeminy, couplets, triplets [salvos], or the R on T phenomenon)
11. Atrial fibrillation or flutter
12. Supine (after patient has been supine for 5 minutes) systolic BP > 160 mm Hg or < 90 mm Hg or diastolic BP > 100 mm Hg or any systolic or diastolic BP that is symptomatic or clinically significant based on the opinion of the Principal Investigator
13. Patients who are receiving warfarin

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Severity of depressive episodes measured using the Montgomery-Asberg Depression Rating Scale (MADRS) | Baseline-Week 10

CONTACTS AND LOCATIONS:
Overall Officials: Rajnish Mago, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States